CLINICAL TRIAL: NCT00273897
Title: Direct Current Brain Polarization for Apraxia in Corticobasal Syndrome
Brief Title: Electrical Polarization of the Brain in Corticobasal Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Eric M. Wassermann, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060067; 06-N-0067
Record Dates: First submitted 2006-01-07; First posted 2006-01-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-16

CONDITIONS: Corticobasal Syndrome
Keywords: Dementia Treatment; Hand Function; Clinical Trials; Dementia; Cortical Syndrome; CBS; Apraxia
MeSH Terms: conditions — Corticobasal Degeneration; Dementia; Apraxias

INTERVENTIONS:
Device: Phoresor II

SUMMARY:
This study will test whether DC electrical polarization of the brain can temporarily improve hand function in patients with corticobasal syndrome (CBS). In this degenerative disorder of the brain, nerve cells die over time, causing a progressive decline in the patient's ability to use their hands. This is always worse on one side. Other symptoms include arm or leg stiffness, tremor, gait unsteadiness, and speech difficulty. Some patients also have some decline in thinking ability, such as loss of skilled activities, poor problem solving abilities poor concentration, problems with language, and forgetfulness,. DC electrical polarization of the brain involves placing sponge electrodes on the head and passing a very weak current between them. DC polarization can temporarily improve the ability of healthy people to make word lists and may improve symptoms in some brain diseases.

Patients 40 and older with CBS who have participated in NINDS protocol 02-N-0001 ("Testing a Model of the Representational Knowledge Stored in the Human Prefrontal Cortex") may be eligible for this study. In protocol 02-N-0001, participants provide a medical history, undergo a neurological examination, PET scanning and MRI, and complete tests, such as sitting in front of a computer monitor and press a key to indicate a decision about what appears on the screen (for example, whether a statement is accurate) and answering questions from a test examiner.

For the current protocol, participants have three 2-hour testing sessions at the NIH Clinical Center, scheduled at least one day apart. In each session, sponge electrodes are placed on the head so that they affect different areas of the brain. Two areas are involved with hand movement; the third does not. The electrodes are dampened with water and attached to the sides of the patient's head. When the current is turned on, the patient may feel some tingling. The current is on for 40 minutes, but can be reduced or stopped early if the tingling becomes uncomfortable.

Before and during each session, the patients' hand function is tested by having them perform and imitate some actions, insert pegs into holes on a board, and tap their index finger as fast as they can. Part or all of the sessions are videotaped for use in evaluating the effects of DC polarization.

DETAILED DESCRIPTION:
Objective: In a recent sham-controlled pilot study, we showed that surface anodal direct current (DC) polarization can improve verbal fluency in frontotemporal dementia patients. Corticobasilar syndrome is a related disorder that presents with disordered limb movement, particularly the loss of stored motor programs, (ideational/ideomotor apraxia) and impaired hand function. Conventional neurorehabilitation is typically unsuccessful in this disorder. We wish to see whether anodal polarization of the inferior parietal cortex (IPC) in CBS patients leads to improved movement and whether the improvement is specifically in the generation of stored movements (praxis). We will also apply polarization to the primary sensorimotor area (SM1), where we expect any effects to be on elemental aspects of movement, such as finger tapping speed. Study population: Twenty CBS patients will be enrolled. Design: This single blind crossover study will have three arms: anodal DC to IPC, anodal DC to SM1, and a control condition: polarization with the electrodes placed on the right and left occipital areas. Outcome Measures: The primary outcome measure is a validated test of ideational and ideomotor apraxia. Secondary outcomes are measures of hand dexterity and coordination.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinically diagnosed CBS, consisting of progressive asymmetric rigidity and apraxia and additional findings suggesting cortical (e.g., one or more of the following: alien limb phenomenon, apraxia of speech, cortical sensory loss, constructional dyspraxia, hemisensory neglect, myoclonus, mirror movements) and basal ganglionic (e.g., one or more of the following: bradykinesia, dystonia, tremor, postural instability) dysfunction.
* Patients fitting these criteria will be identified among those referred to protocol 02-N-0001. All must have been evaluated under this protocol.
* Enough residual hand function on one side to perform the tests.
* Age greater than or equal to 40: This limit is justified because the diagnosis of CBS would be very uncertain in anyone under this age.

EXCLUSION CRITERIA:

* Presence of metal in the cranial cavity or calvarium.
* Uncontrolled medical problems, such as uncontrolled diabetes mellitus, hypertension, airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for participation.
* Broken skin in the area of the electrodes.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-12-30; Primary Completion 2007-12-11 (Actual)

PRIMARY OUTCOMES:
Validated test of ideational and ideomotor apraxia.

SECONDARY OUTCOMES:
Measures of hand dexterity and coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boeve BF, Lang AE, Litvan I. Corticobasal degeneration and its relationship to progressive supranuclear palsy and frontotemporal dementia. Ann Neurol. 2003;54 Suppl 5:S15-9. doi: 10.1002/ana.10570. No abstract available. PMID 12833363
- [Background] Boeve BF, Maraganore DM, Parisi JE, Ahlskog JE, Graff-Radford N, Caselli RJ, Dickson DW, Kokmen E, Petersen RC. Pathologic heterogeneity in clinically diagnosed corticobasal degeneration. Neurology. 1999 Sep 11;53(4):795-800. doi: 10.1212/wnl.53.4.795. PMID 10489043
- [Background] Herwig U, Satrapi P, Schonfeldt-Lecuona C. Using the international 10-20 EEG system for positioning of transcranial magnetic stimulation. Brain Topogr. 2003 Winter;16(2):95-9. doi: 10.1023/b:brat.0000006333.93597.9d. PMID 14977202